CLINICAL TRIAL: NCT04239014
Title: A Phase 2 Randomized, Multi-Centre Study to Investigate the Efficacy and Tolerability of a Second Maintenance Treatment in Patients With Platinum Sensitive Relapsed Epithelial Ovarian Cancer, Who Have Previously Received PARP Inhibitor Maintenance Treatment
Brief Title: A Study to Evaluate the Effectiveness and Tolerability of a Second Maintenance Treatment in Participants With Ovarian Cancer, Who Have Previously Received Polyadenosine 5'Diphosphoribose [Poly (ADP Ribose)] Polymerase Inhibitor (PARPi) Treatment.
Acronym: DUETTE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor made the decision to terminate the DUETTE study based on the interim analysis of the VIOLETTE study (NCT03330847) investigating the combination of ceralasertib and Olaparib, where study closure was recommended due to insufficient efficacy.
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6018C00004
Record Dates: First submitted 2020-01-21; First posted 2020-01-23 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Ovarian Cancer
Keywords: Platinum Sensitive Relapsed Epithelial Ovarian Cancer; Polyadenosine 5'diphosphoribose (poly [ADP ribose]) polymerase inhibitor (PARPi)
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib; ceralasertib

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The olaparib and placebo arms will be double blinded, whereas the ceralasertib+olaparib arm will be open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (ceralasertib+olaparib) (Experimental): Participants received ceralasertib 160 mg QD PO on Days 1 to 7 plus olaparib 300 mg BD PO continuous (28 day cycle).
  Interventions: Drug: Olaparib; Drug: Ceralasertib
- Arm 2 (olaparib monotherapy) (Experimental): Olaparib 300 mg BD PO daily continuous.
  Interventions: Drug: Olaparib
- Arm 3 (placebo) (Experimental): Placebo to match olaparib BD PO daily continuous.
  Interventions: Drug: Placebo to match olaparib

INTERVENTIONS:
Drug: Olaparib — Olaparib 300 mg BD (2 × 150 mg tablets) continually in the olaparib monotherapy and ceralasertib+olaparib treatment arms.
  Other Names: AZD2281
  Arms: Arm 1 (ceralasertib+olaparib); Arm 2 (olaparib monotherapy)
Drug: Ceralasertib — Ceralasertib 160 mg QD (2 × 80 mg tablets) from Days 1 to 7 (inclusive) of every 28-day cycle.
  Other Names: AZD6738
  Arms: Arm 1 (ceralasertib+olaparib)
Drug: Placebo to match olaparib — Per olaparib
  Arms: Arm 3 (placebo)

SUMMARY:
To investigate the effectiveness and tolerability of a second maintenance treatment in participants with platinum-sensitivity relapsed (PSR) epithelial ovarian cancer, who have previously received PARPi maintenance treatment and who have benefit (complete response [CR] or partial response [PR]) or stable disease (SD) from further platinum based chemotherapy.

DETAILED DESCRIPTION:
This is a Phase II, randomised, multicentre study to investigate the efficacy and tolerability of a second maintenance treatment in participants with PSR epithelial ovarian cancer, who have previously received PARPi maintenance treatment and who have benefit (CR or PR) or SD from further platinum based chemotherapy.

Participants will be recruited globally from approximately 120 study sites in the USA, Canada, Middle East and Europe.

Approximately 192 participants fulfilling all of the inclusion criteria and none of the exclusion criteria will be randomised in a 1:1:1 ratio to the following 3 treatment arms (64 participants per arm):

* Arm 1 (ceralasertib+olaparib): Ceralasertib 160 mg once daily (QD) orally or per os (PO) on Days 1 to 7 plus olaparib 300 mg twice daily (BD) PO continuous (28 day cycle)
* Arm 2 (olaparib monotherapy): Olaparib 300 mg BD PO daily continuous
* Arm 3 (placebo): Placebo to match olaparib BD PO daily continuous

The olaparib and placebo arms will be double blinded, whereas the ceralasertib+olaparib arm will be open label. It is expected that approximately 320 participants will be screened.

The study achieved First Subject In date, but enrollment equals 0 as 7 participants have signed the Informed Consent Form (ICF) and were later screen failed.

ELIGIBILITY:
Inclusion Criteria:

* Capable of providing signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in the Clinical Study Protocol (CSP).
* Provision of signed and dated, written ICF prior to any mandatory study specific procedures, sampling, and analyses.
* Female ≥18 years of age at the time of signing the ICF.
* Eastern Cooperative Oncology Group performance status 0 to 1 within 28 days of randomization.
* Participants with relapsed histologically confirmed diagnosis of high grade epithelial ovarian cancer (including primary peritoneal and/or fallopian tube cancer), with disease relapse on or after completion of PARPi maintenance therapy and who have not received any intervening systemic treatment since discontinuation of PARPi (this excludes the platinum based chemotherapy received during Screening Part 1 of this study).
* A minimum of 6 months of prior PARPi treatment received in the maintenance setting for PSR ovarian cancer (a minimum of 12 months is required if the participant received PARPi maintenance following first line chemotherapy). If the prior PARPi used was olaparib then participants must have received treatment without significant toxicity or the need for a permanent dose reduction.
* Disease relapse in the second line (first relapse) or third line (second relapse) setting.
* Able to provide and consent to the collection of a contemporaneous tumor tissue biopsy and blood sample.
* Able to provide a Formalin Fixed Paraffin Embedded archival tumour tissue block from the time of primary tumour diagnosis (taken ideally prior to receiving any systemic treatment, and definitely prior to first PARPi treatment) for prospective Breast cancer susceptibility gene (BRCA) status testing. If tumour blocks are unavailable, tissue sections are acceptable with a minimum requirement of at least 20 unstained sections on uncharged slides without cover slips. Fine needle aspirates are not acceptable.
* Where the patient has previously been tested for germline or somatic BRCA alterations using a verified and well-validated test in line with local regulations, performed in a locally accredited laboratory (eg, College of American Pathologists/Clinical Laboratory Improvement Amendments laboratory, where available), and signed consent to provide a copy of the BRCA report.
* Platinum-sensitive disease at the time of disease relapse, i.e, platinum-treatment free survival of greater than 6 months as defined by the Gynecological Cancer Intergroup (Wilson et al 2017).
* For the platinum-based chemotherapy course received following pre screening (Part 1) and prior to entering the main screening (Part 2).
* Any prior palliative radiation must have been completed at least 7 days prior to the start of study drugs, and participants must have recovered from any acute adverse effects prior to the start of study treatment.
* Normal organ and bone marrow function measured within 28 days prior to randomization.
* Participant is willing and able to comply with the CSP for the duration of the study including undergoing treatment and scheduled visits and examinations.
* Participants must have a life expectancy of ≥16 weeks.
* Participants must be able to swallow tablets whole.
* For inclusion in the optional (deoxyribonucleic acid) genetics research, study participants must fulfil the following criterion:

Provide informed consent for the genetic sampling and analyses. If a participant declines to participate in the genetics research, there will be no penalty or loss of benefit to the participant. A participant who declines genetics research participation will not be excluded from any other aspect of the main study.

* Participant's body weight must be >30 kg.
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential.
* Women of childbearing potential and their partners, who are sexually active, must agree to the use of 2 highly effective forms of contraception in combination from the signing of the informed consent (Screening Part 1), throughout the period of taking study treatment and for at least 6 months after the last dose of study drug(s).

Exclusion Criteria:

* Participants who have had drainage of their ascites during the final 2 cycles of their last chemotherapy regimen or during the period between completion of chemotherapy and first dose of study treatment.
* Participants with current signs or symptoms of bowel obstruction, including sub-occlusive disease, related to underlying disease.
* History of leptomeningeal carcinomatosis.
* Participants with symptomatic uncontrolled brain metastases.

  1. A scan to confirm the absence of brain metastases is not required.
  2. Participants whose brain metastases have been treated may participate provided they show radiographic stability. In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved or be stable (Common Terminology Criteria for Adverse Events [CTCAE] Grade <2) either, without the use of steroids, or are stable on a steroid dose of ≤10 mg/day of prednisone or its equivalent and stable on anti convulsants if required for at least 14 days prior to the start of treatment.
  3. Participants with spinal cord compression are not eligible unless considered to have received definitive treatment for this and have evidence of clinically SD for >28 days and have not received steroid treatment for at least 14 days prior to the start of study treatment.
* History of another primary malignancy except for:

  1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence;
  2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease;
  3. Adequately treated carcinoma in situ without evidence of disease.
* Major surgical procedures (as defined by the investigator) ≤28 days of beginning study treatment, or minor surgical procedures ≤7 days. No waiting period required following port a cath or other central venous access placement.
* Persistent toxicities (≥CTCAE Grade 2) caused by previous cancer therapy, excluding alopecia and CTCAE Grade 2 peripheral neuropathy. Note: participants with signs of ongoing complications from radiation therapy are not eligible for this study.
* Participants with myelodysplastic syndrome (MDS) /acute myeloid leukemia (AML) or with features suggestive of MDS/AML.
* Resting electrocardiogram indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator, or participants with congenital long QT syndrome.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* History of allogeneic organ transplantation including previous allogeneic bone marrow transplant or double umbilical cord blood transplantation.
* History of active primary immunodeficiency.
* Active infection including tuberculosis (TB), hepatitis B (known positive hepatitis B virus [HBV] surface antigen [HBsAg] result), hepatitis C (HCV), or human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies). Participants with a past or resolved HBV infection are eligible. Participants positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid.
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, active interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations.
* Current dependency on total parenteral nutrition or intravenous (iv) fluid hydration.
* Whole blood transfusions in the last 120 days prior to entry to the study.
* Cytotoxic chemotherapy, hormonal or non hormonal targeted therapy within 21 days of Cycle 1, Day 1 is not permitted. The participant can receive a stable dose of bisphosphonates or denosumab for bone metastases, before and during the study as long as these were started at least 5 days prior to study treatment.
* Participation in another clinical study with an IP during the chemotherapy course immediately prior to randomisation or during the course of the study.
* Previous treatment with ceralasertib or other ataxia telangiectasia and Rad3-related protein, Checkpoint kinase 1 or deoxyribonucleic acid damage response inhibitor (excluding PARPi).
* Exposure to a small molecule IP within 30 days or 5 half-lives (whichever is longer) prior to randomization. The minimum washout period for immunotherapy and bevacizumab shall be 42 days.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study treatment.
* Concomitant use of known strong cytochrome P450 (CYP) 3A inhibitors or moderate CYP3A inhibitors. The required washout period prior to starting study treatment is 2 weeks.
* Concomitant use of known strong CYP3A inducers or moderate CYP3A inducers. The required washout period prior to starting study treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Involvement in the planning and/or conduct of the study (applies to Sponsor staff and/or staff at the study site).
* Previous randomization in the present study.
* Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions and requirements.
* Pregnant or lactating women.

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female ≥18 years of age at the time of signing the informed consent form (ICF).
Enrollment: 0 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | To assess from the time of randomization until the date of objective disease progression or death (by any cause in the absence of progression) or approximately up to 2.5 years.
  To assess the efficacy of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.

SECONDARY OUTCOMES:
Overall survival (OS) | To assess every 8 weeks (±7 days) for first 72 weeks following objective disease progression or treatment discontinuation and then every 12 weeks, up to approximately 2.5 years.
  To further assess the efficacy of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo; and to assess the efficacy of maintenance ceralasertib+olaparib combination therapy compared with olaparib monotherapy.
Time to second progression | To assess every 8 weeks (±7 days) for first 72 weeks following objective disease progression or treatment discontinuation and then every 12 weeks, up to approximately 2.5 years.
  To further assess the efficacy of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo; and to assess the efficacy of maintenance ceralasertib+olaparib combination therapy compared with olaparib monotherapy. A participant's second progression status is defined according to the local standard clinical practice and may involve any of; investigator assessment of radiological progression, cancer antigen 125 (CA 125) progression, symptomatic progression or death.
Objective response rate | At baseline, every 8 weeks for first 72 weeks, then every 12 weeks after randomization until objective disease progression or approximately up to 2.5 years.
  To further assess the efficacy of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo; and to assess the efficacy of maintenance ceralasertib+olaparib combination therapy compared with olaparib monotherapy.
Duration of response | At baseline, every 8 weeks for first 72 weeks, then every 12 weeks after randomization until objective disease progression or approximately up to 2.5 years.
  To further assess the efficacy of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo; and to assess the efficacy of maintenance ceralasertib+olaparib combination therapy compared with olaparib monotherapy.
Percentage change in tumour size | At baseline, every 8 weeks for first 72 weeks, then every 12 weeks after randomization until objective disease progression or approximately up to 2.5 years.
  To further assess the efficacy of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Plasma concentration data for olaparib and ceralasertib | At cycle 1 Day 1 and Day 7
  To evaluate the pharmacokinetic (PK) exposure of ceralasertib+olaparib combination therapy.
Change from baseline in European Organisation for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC-QLQ) C30 | At Cycle1 Day 1, every 4 weeks from Cycle 1 Day 1 until treatment discontinuation, and follow-up 30 days after last dose of study medication.
  To assess the impact of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo on participants' symptoms, functioning, and Health-related quality of life (HRQoL). Questions are grouped into functional scales, symptom scales, a global health status / quality of life (QoL) scale, assessing additional symptoms commonly reported by cancer participants, and the financial impact of the disease. All but 2 questions are rated on a 4 point verbal rating scale: "Not at all," "A little," "Quite a bit," and "Very much." The 2 questions concerning global health status and QoL have 7 point scales with ratings ranging from "Very poor" to "Excellent." For each of the 15 domains, final scores are transformed such that they range from 0 to 100, where higher scores indicate better functioning, better QoL, or worse symptoms.
Change from baseline in EORTC-QLQ-OV28 | At Cycle1 Day 1, every 4 weeks from Cycle 1 Day 1 until treatment discontinuation, and follow-up 30 days after last dose of study medication.
  To assess the impact of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo on participants' symptoms, functioning, and HRQoL It consists of 28 items assessing abdominal/gastrointestinal symptoms (6 items), peripheral neuropathy (2 items), other chemotherapy side effects (5 items), hormonal symptoms (2 items), body image (2 items), attitudes to disease/treatment (3 items), sexuality (4 items) and 4 other single items. All questions are rated on a 4 point verbal rating scale: "Not at all," "A little," "Quite a bit," and "Very much." Final scores are transformed such that they range from 0 to 100, where higher scores indicate greater functioning, greater QoL, or greater level of symptoms.
Time to earliest progression by RECIST 1.1 or CA-125 or death | At baseline, every 8 weeks for first 72 weeks, then every 12 weeks after randomization until objective disease progression or approximately up to 2.5 years.
  Time to progression by RECIST 1.1 or CA-125 progression or death is defined as the time from randomisation to the earlier date of RECIST 1.1 or CA-125 progression or death by any cause.

OTHER OUTCOMES:
Number of participants with adverse events (AEs) | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal physical examination | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal Eastern Cooperative Oncology Group (ECOG) performance status (PS) | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number participants with abnormal systolic and diastolic blood pressure | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal pulse | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal body temperature | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal electrocardiogram | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal hemoglobin (Hb) | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal leukocyte count | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal absolute neutrophil count (ANC) | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal absolute lymphocyte count | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal platelet count | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal mean cell volume | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal serum creatinine | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal serum total bilirubin | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal serum alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal serum potassium, calcium and sodium | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal plasma glucose | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal serum lactate dehydrogenase | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal creatinine clearance | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal serum urea or blood urea nitrogen | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal plasma total protein | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal urine Hb/erythrocytes/blood | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal urine protein/albumin | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal urine glucose | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal urine ketones | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal urine pH | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal specific gravity | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
Number of participants with abnormal urine bilirubin | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess the safety and tolerability of maintenance olaparib monotherapy and ceralasertib+olaparib combination therapy compared with placebo.
European quality of life 5 dimensions, 5 level | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess both European quality of life descriptive system and European quality of life visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The participant is asked to indicate his health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the participant's health state.
  The EQ VAS records the participant's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'the best health you can imagine' and 'the worst health you can imagine'.
Patient Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess tolerability from the participants perspective. PRO-CTCAE is an item library of symptomatic AEs experienced by patients while undergoing treatment of their cancer. PRO questionnaires completed at site visits must be completed prior to treatment administration
Patient global impression of severity | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess overall severity of participant's cancer symptoms over the past week. The item is rated using a 6 point verbal rating scale from "No Symptoms" to "Very Severe".
Patient global impression of change | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To assess overall change in health condition since the start of study treatment(s). The item is rated using a 7 point Likert type scale from "Much Better" to "Much Worse".
Patient global impression-treatment tolerability | From Cycle 1 Day 1 to follow-up 30 days after the last dose of study medication.
  To asses overall bother associated with symptomatic AEs. The item is rated using a 6 point verbal scale from "Not at All" to "Very Much".
Patient global impression-benefit risk | From Cycle 1 Day 1 to 12 weeks and 16 weeks of study medication.
  To asses the participant's perception of the overall benefits and risks of treatment. The 5 items to be assessed included overall trial experience, efficacy, side effects, convenience, and overall assessment of the benefits and harms of treatment. Items are rated on 5 or 6 point verbal rating or Likert type scales.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Amit Oza, MD (Lon) FRCP FRCPC, Principal Investigator — Princess Margaret Cancer Centre, UHN and Mt. Sinai Health System
Locations (25):
- United States (21):
  - Research Site, Anchorage, Alaska
  - Research Site, La Jolla, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, West Hollywood, California
  - Research Site, Hartford, Connecticut
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Louisville, Kentucky
  - Research Site, Covington, Louisiana
  - Research Site, Florham Park, New Jersey
  - Research Site, Teaneck, New Jersey
  - Research Site, Cleveland, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Abington, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Houston, Texas
  - Research Site, Seattle, Washington
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Research Site, Napoli, Italy
- Research Site, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please re-refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] McMullen M, Karakasis K, Loembe B, Dean E, Parr G, Oza AM. DUETTE: a phase II randomized, multicenter study to investigate the efficacy and tolerability of a second maintenance treatment in patients with platinum-sensitive relapsed epithelial ovarian cancer, who have previously received poly(ADP-ribose) polymerase (PARP) inhibitor maintenance treatment. Int J Gynecol Cancer. 2020 Nov;30(11):1824-1828. doi: 10.1136/ijgc-2020-001694. Epub 2020 Sep 2. PMID 32878963